CLINICAL TRIAL: NCT02279940
Title: Rivaroxaban Acute Stroke Safety Study
Acronym: RASS
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Ken Butcher, Assistant Professor, University of Alberta
Other Study IDs: Version 1.0
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Acute Ischemic Stroke; Transient Ischemic Attack
Keywords: rivaroxaban; stroke; transient ischemic attack; ischemia
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Stroke; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
Atrial fibrillation is a common cardiac arrhythmia and a major risk for ischemic stroke. Furthermore the risk of stroke is higher in the first month after transient ischemic attack (TIA)/stroke. Rivaroxaban has been approved by Health Canada over period of last two years for prevention of stroke and have been found equally effective as oral Vitamin K antagonist. The foremost benefits of NOAC are reduced intracranial bleeding risk and does not require coagulation monitoring.

Optimal timing of anticoagulation after TIA/stroke in patients with known non-valvular atrial fibrillation is not known. The practice is variable and opinion based. The bias for many stroke physicians and neurologists is to start later (after 1-2weeks) to prevent hemorrhagic transformation thus possibly exposing the patients to an increased risk of recurrence. The product monograph for the drug suggest to wait for variable of 3 to 14 days before starting the NOAC (Waiting period:14 days for dabigatran and rivaroxaban, 7 days for Apixaban after ischemic stroke and three days after TIA for rivaroxaban). The times have been chosen arbitrary.

The investigators aim to study incidence of symptomatic hemorrhage in patients with non-valvular atrial fibrillation who are initiated with new oral anticoagulants early after TIA and stroke.

DETAILED DESCRIPTION:
Background:

It is clearly established that patients with atrial fibrillation who have suffered a stroke/TIA are at high risk for recurrence and require long-term anticoagulation. What is unknown is the optimal timing of anticoagulation after an ischemic stroke has occurred. Following cardioembolic stroke, atrial fibrillation patients are at risk for early recurrent thrombo-embolism. Estimates of the rate of recurrent stroke in this setting vary widely. Previous studies have indicated new ischemic strokes occur at rates anywhere from 3% to 20% within two weeks of the index event. This is the primary rationale for early anticoagulation after cardioembolic stroke. There is some evidence that early anticoagulation is associated with improved outcomes after ischemic stroke. Indeed, it has been shown that early heparin use does reduce recurrent ischemic stroke risk by 2.1%, but this is offset by a 1.7% increase in the rate of HT. Studies of low molecular weight and unfractionated heparin use in acute stroke have generally indicated these agents are associated with moderately increased risk of HT. There are currently no data indicating the frequency of HT associated with early warfarin treatment, without heparin bridging.

Based on the above evidence, current best practice guidelines recommend against urgent anticoagulation in patients with moderate to severe ischemic stroke, however, due to the elevated risk of hemorrhagic transformation (HT) immediately after stroke. A specific time point at which to begin anticoagulation is not recommended in guideline statements. This clinical equipoise has resulted in significant variation in practice patterns. Currently, most CSC physicians base the timing of anticoagulation on clinical severity and infarct size, as seen on CT scan. Most physicians will defer anticoagulation anywhere from 5 to 14 days after ischemic stroke when infarct volume is extensive. In patients with small infarct volumes, assessed with CT or MRI, however, anticoagulation is often begun within 24-72 hours of stroke onset, and in some cases immediately after clinical assessment and CT scan.

Currently, Bayer has no data related to early use of rivaroxaban after TIA or ischemic stroke. Although a randomized study of delayed versus early anticoagulation with rivaroxaban will ideally answer this question, at the moment, there is no feasibility or safety data. There is also insufficient data in the present literature to indicate what the true event rates for both symptomatic hemorrhagic transformation and recurrent cerebral ischemia are. These data can be obtained by prospectively collecting clinical and imaging data from patients who are treated, as per standard clinical practice in most Canadian stroke centres, within this 14-day period of clinical uncertainty. The results of this registry will be used to assess the safety and feasibility of a larger randomized controlled trial of early versus delayed rivaroxaban use after stroke/TIA.

Study Design:

The Rivaroxaban Acute Stroke Safety Study (RASS) is an investigator initiated multi-center, prospective, open label, single arm phase IV study.

Objectives and Hypothesis:

The primary aim of the Rivaroxaban Acute Stroke Study registry is to demonstrate the safety of early anticoagulation with rivaroxaban following cardioembolic stroke and TIA. Safety will be established by demonstrating low rates of hemorrhage in this setting. The secondary study objective is to document the rate of recurrent cerebrovascular ischemic events. It is fully recognized that this uncontrolled registry study is not properly designed and under-powered to demonstrate a reduction in cerebrovascular ischemic events. The investigators hypothesize that early initiation of rivaroxaban within the first 14 days of stroke or TIA is not associated with increased symptomatic intracranial haemorrhage.

Baseline Data (within 14 days of TIA/minor stroke):

Standard clinical assessments and data will be collected. This will include baseline National Institutes of Health Stroke Scale NIHSS, Glasgow Coma Scale (GCS), Montreal Cognitive Score (MoCA) and vital signs, which will be recorded in a case report form. Stroke risk factors, past medical history and medications, baseline complete blood count, coagulation profile and renal function tests will also be recorded.

Treatment:

Patients will be treated with rivaroxaban within 14 days of symptom onset according to the practice pattern of the attending stroke physician. The study participation would be considered after patient has been initiated on Rivaroxaban. The dose of rivaroxaban will be determined by age and renal function. Patients >80 years old and/or with GFR 30-50 ml/min will receive 15 mg qd, and all other patients will receive 20 mg qd. The study team members would then approach the patients for possible recruitment in the study after obtaining informed consent.

Imaging Procedures:

Acute baseline CT scans will be collected (standard of care). All patients will have MRI including susceptibility weighted imaging after recruitment within the first 24 hours and a follow-up MRI scan 7±2 days after enrolment, in order to assess for early asymptomatic hemorrhagic transformation. In the event of any clinical deterioration, a repeat CT scan will be performed immediately. The investigators hypothesize micro-hemorrhages may predict symptomatic bleeding. In addition, any supplemental brain imaging completed within the first 30 days after enrolment will be collected.

Clinical Follow-up Assessments:

All patients will be followed for 90 days. This is the standard post-stroke assessment period (the majority of neurological and functional recovery occurs within this time frame). Patients will be assessed clinically at Day 1, Day 7, and Day 90. At each visit, patients will again be examined by a stroke Fellow and/or Neurologist. On each visit, vital signs will be noted, a comprehensive neurologic examination will be performed and mRS and NIHSS will be recorded. Patients will be interviewed in detail to identify and ascertain any recurrent vascular event suggestive of a stroke or TIA. Work-up to determine the underlying etiology of stroke will be reviewed and any change in management plan will be recorded.

Statistical Analysis Plan and Power Calculation:

The primary outcome will be tested with a single sample t-test. The null hypothesis is that the frequency of symptomatic hemorrhagic transformation is <2%. A convenience sample of 50 patients is planned initially. This will provide initial safety and feasibility data that can be used to plan future definitive studies as required. The primary efficacy analysis will be on an intention-to-treat basis.

Data Safety Monitoring and Adverse Event Reporting:

Investigators will report serious adverse events (SAE), using standardized event, resolution and association codes. The SAE reporting period includes the entire treatment duration and an additional week. All SAEs will be reported. Non-serious Adverse Events (AEs) unrelated to rivaroxaban treatment will not be reported.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be ≥ 18 years of age.
* All patients will have a diagnosis of minor ischemic stroke, defined as NIHSS score ≤ 8, or Transient Ischemic Attack (TIA), defined as acute focal neurological deficits, with complete resolution of symptoms within 24 h of onset. In cases where onset time cannot be established, it will be considered to be the time when the patient was last known to be well.
* Atrial Fibrillation (AF, paroxysmal or persistent). AF must be confirmed with ECG/Holter monitor, or by history (clinical documentation of previous AF must be provided).
* All included patients will be prescribed rivaroxaban following their stroke/TIA.

Exclusion Criteria:

* Acute or chronic renal failure, defined as eGFR <30 ml/min (Cockcroft Gault formula).
* Known hypersensitivity to rivaroxaban.
* Prior treatment with rivaroxaban or any other novel oral anticoagulant (including all Factor Xa antagonists). Treatment with warfarin prior to the stroke/TIA is acceptable, but enrolment cannot begin until the INR is ≤2.0.
* Any significant ongoing systemic bleeding risk, i.e. active GI/GU bleeding or recent major surgery.
* Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
* Recent past history or clinical presentation of ICH, subarachnoid haemorrhage (SAH), arterio-venous (AV) malformation, aneurysm, or cerebral neoplasm. At the discretion of each Investigator.
* Hereditary or acquired haemorrhagic diathesis.
* Stroke mimics (such as seizures, migraine etc.)
* Contraindications to MRI will also be excluded, including metallic implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with atrial fibrillation (new onset or previous history) with acute ischemic stroke or TIA will be screened from Emergency Department or stroke unit. A total of 50 male and female patients will be recruited within 24 hours of symptom onset. Informed consent will be obtained from the patient or substitute decision maker, in all cases prior to enrolment.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Symptomatic Hemorrhagic Transformation Rate | 30 days post-treatment
  PH2 associated with clinical deterioration, defined as worsening of NIHSS score of 4 or more points within 30 days of initiating anticoagulant therapy

SECONDARY OUTCOMES:
Any parenchymal haemorrhage (PH1 or PH2) on follow-up MRI scan at 7±2 days post-enrolment. | 7 days post-treatment
Recurrent Transient Ischemic Attack/Ischemic Stroke within 90 days of enrolment. | 90 days following enrollment
Systemic hemorrhagic complication rate within 90 days of enrolment. | 90 days following enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada